CLINICAL TRIAL: NCT04220840
Title: The Damage Control Strategy for the Treatment of Perforated Diverticulitis of the Sigmoid Colon With Diffuse Peritonitis - a Retrospective, Multicenter, Transnational Cohort Study
Brief Title: The Damage Control Strategy for the Treatment of Perforated Diverticulitis of the Sigmoid Colon With Diffuse Peritonitis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Städtisches Klinikum München GmbH (Other)
Collaborators: Charite University, Berlin, Germany (Other); Medical University Innsbruck (Other); University of Pisa (Other); Cardarelli Hospital (Other)
Responsible Party: Principal Investigator, Dr. Maximilian Sohn, M.D., Dr. med., Attending Surgeon, Städtisches Klinikum München GmbH
Other Study IDs: DCS-INT-2020
Record Dates: First submitted 2020-01-03; First posted 2020-01-07 (Actual); Last update posted 2023-09-08 (Actual); Status verified 2023-09

CONDITIONS: Perforated Diverticulitis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Study Group: All consecutive patients who underwent damage control surgery (DCS) for perforated diverticulitis of the sigmoid colon with generalized Peritonitis in one of the participating centers
  Interventions: Procedure: Damage control strategy
- Control group: All consecutive patients who underwent other than DCS surgery (resection with primary anastomosis, Hartmann´s procedure, laparoscopic lavage) for perforated diverticulitis of the sigmoid colon with generalized Peritonitis in one of the participating centers which do not apply DCS routinely.
  Interventions: Procedure: Damage control strategy

INTERVENTIONS:
Procedure: Damage control strategy — The damage control strategy constitutes a two stage procedure.
  Emergency surgery:
  limited resection oft he diseased colonic segment with oral and aboral blind closure, abdominal lavage, temporary vacuum assisted abdominal closure
  Second look surgery (48-72 hours later):
  reexploration with
  1. definite reconstruction (Colorectal anastomosis -/+ diverting ileostomy vs. end colostomy)
  2. lavage, vacuum assisted abdominal closure, third look 72 hours after emergency surgery

SUMMARY:
The best approach for the treatment of perforated diverticulitis of the sigmoid colon is still under debate. Concurrent techniques are 1) resection with primary colorectal anastomosis with or without additional loop ileostomy; 2) end colostomy (Hartmann´s procedure); 3) Damage control strategy; 4) laparoscopic lavage and placement of a drainage. It is hypothesized, that the use of the damage control strategy leads to a significant reduction of the stoma rate.

The damage control strategy constitutes a two stage procedure.

Emergency surgery:

limited resection of the diseased colonic segment with oral and aboral blind closure, abdominal lavage, temporary vacuum assisted abdominal closure

Second look surgery (48-72 hours later):

Reexploration with

1. definite reconstruction (Colorectal anastomosis -/+ diverting ileostomy vs. end colostomy)
2. lavage, vacuum assisted abdominal closure, third look 72 hours after emergency surgery

Within the study, data of DCS-procedures will be collected retrospectively in a multicentric and transnational approach. Those will be compared to a cohort of patients treated with a "no-DCS"-technique (resection with primary anastomosis or Hartmann´s procedure).

DETAILED DESCRIPTION:
Research question/objective of the study

It is assumed that the application of the Damage Control Strategy (DCS) in patients with perforated diverticulitis of the sigmoid colon with generalized peritonitis leads to a reduction of the stoma rate with the same degree of safety as other procedures (Hartmann´ procedure, sigmoid resection with primary anastomosis, laparoscopic lavage).

Definitions

The damage control strategy constitutes a two stage procedure.

Emergency surgery:

limited resection of the diseased colonic segment with oral and aboral blind closure, abdominal lavage, temporary vacuum assisted abdominal closure

Second look surgery (48-72 hours later):

Reexploration with

1. definite reconstruction (Colorectal anastomosis -/+ diverting ileostomy vs. end colostomy)
2. lavage, vacuum assisted abdominal closure, third look 72 hours after emergency surgery

Basis and scientific knowledge

The majority of patients with acute diverticulitis of the left colon are currently treated conservatively. However, diverticular perforation with diffuse peritonitis remains a challenging and life-threatening situation requiring emergency surgical intervention. Regardless of the frequency and severity of the disease, there is yet no generally accepted treatment algorithm. Sigmoid resection with blind closure of the rectal stump and formation of an end colostomy (Hartmann´s procedure) as well as sigmoid resection with primary anastomosis with or without additional loop ileostomy are alternative procedures. As an additional approach, laparoscopic lavage and drainage has not yet been widely established. Accordingly, the technique is not recommended in the current German S2K guidelines for the treatment of diverticular disease. Within Damage Control Strategy (DCS), a limited resection of the affected sigmoid segment with oral and aboral blind closure is performed during the initial intervention. After abdominal lavage, a temporary vacuum-assisted closure of the abdominal cavity is then performed. 24 to 72 hours later, the decision on the definite reconstruction procedure is made within the scope of the planned second-look laparotomy. Generally, a colorectal anastomosis with or without loop ileostomy is intended. If this is not possible, end colostomy is available as additional option. Principal criteria for the decision on the type of definite reconstruction are the local and general findings of the patient. According to the results of a first cohort from the Innsbruck University Hospital, a colorectal anastomosis can be achieved in almost 80% of patients within second operation. In about half of the patients, a loop ileostomy is additionally created. Using DCS, morbidity and mortality are comparable to the above mentioned competing procedures. An own study from 2016 shows similar results. After the initial hospital stay, 47% of the patients were stoma carriers after the application of DCS, compared to 83% of the patients from the control group to which all "other" surgical procedures (Hartmann operation, Primary anastomosis with or without loop ileostoma) were assigned. At the end of follow-up, 88% of patients were stoma-free after use of DCS. The mortality rate was 11 percent. A systematic review of the available specific literature on DCS is yet underway. The manuscript is currently undergoing peer review at the World Journal of Gastroenterology. In the course of this process the above mentioned results could be confirmed. A total of eight publications from five study groups were identified (status 11/2019). In 73% of the cases a colorectal anastomosis could be performed during the second-look laparotomy. 15% of the patients additionally received a loop ileostomy. End colostomy (secondary Hartmann´s procedure) was necessary in only 27% of the patients. The cumulative anastomotic leak rate was 13%, surgical morbidity 31% and 30-day mortality was 9%. A stoma rate of 45% at discharge should be emphasized. Thus, the number of patients in whom intestinal continuity could be restored during the initial hospital stay was considerably higher when using the damage control strategy than in most studies on the treatment of perforated diverticulitis with diffuse peritonitis. In addition, a stoma rate of <50% at discharge was achieved. These aspects should be highlighted as key benefits. Further positive aspects of the method are the fast and technically simple focus repair during the initial intervention.

ELIGIBILITY:
Inclusion Criteria:

all patients who were operated for perforated diverticulitis with generalized peritonitis

Exclusion Criteria:

incomplete data sets

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All consecutive patients who underwent surgery for perforated diverticulitis of the sigmoid colon with generalized peritonitis will be included into the analysis
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2020-11-01 (Actual); Primary Completion 2023-12-01 (Estimated); Study Completion 2024-06-01 (Estimated)

PRIMARY OUTCOMES:
Stoma rate at the end of the index hospital stay | 30 days after surgery for definite reconstruction
  rate of enterostomies (Loop ileostomy and end colostomy) at the end of the hospital stay, associated to the emergency operation

SECONDARY OUTCOMES:
Stoma rate over the long term | through study completion, an average of 1 year
  rate of enterostomies (Loop ileostomy and end colostomy) at the end of the follow-up
30-day Morbidity | 30 days after surgery for definite reconstruction
  Morbidity assessed by the Clavien-Dindo classification
30-day Mortality | 30 days after surgery for definite reconstruction
  Mortality

CONTACTS AND LOCATIONS:
Locations (1):
- Dr. Maximilian Sohn, Munich, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Sohn M, Iesalnieks I, Agha A, Steiner P, Hochrein A, Pratschke J, Ritschl P, Aigner F. Perforated Diverticulitis with Generalized Peritonitis: Low Stoma Rate Using a "Damage Control Strategy". World J Surg. 2018 Oct;42(10):3189-3195. doi: 10.1007/s00268-018-4585-y. PMID 29541823
- [Result] Sohn MA, Agha A, Steiner P, Hochrein A, Komm M, Ruppert R, Ritschl P, Aigner F, Iesalnieks I. Damage control surgery in perforated diverticulitis: ongoing peritonitis at second surgery predicts a worse outcome. Int J Colorectal Dis. 2018 Jul;33(7):871-878. doi: 10.1007/s00384-018-3025-7. Epub 2018 Mar 13. PMID 29536238
- [Result] Sohn M, Agha A, Heitland W, Gundling F, Steiner P, Iesalnieks I. Damage control strategy for the treatment of perforated diverticulitis with generalized peritonitis. Tech Coloproctol. 2016 Aug;20(8):577-83. doi: 10.1007/s10151-016-1506-7. Epub 2016 Jul 22. PMID 27448296
- [Result] Kafka-Ritsch R, Birkfellner F, Perathoner A, Raab H, Nehoda H, Pratschke J, Zitt M. Damage control surgery with abdominal vacuum and delayed bowel reconstruction in patients with perforated diverticulitis Hinchey III/IV. J Gastrointest Surg. 2012 Oct;16(10):1915-22. doi: 10.1007/s11605-012-1977-4. Epub 2012 Jul 28. PMID 22843083